CLINICAL TRIAL: NCT02024932
Title: A Two-part Placebo-controlled Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of BVS857 in Patients With Spinal and Bulbar Muscular Atrophy (SBMA)
Brief Title: Safety, Tolerability, and Efficacy of BVS857 in Patients With Spinal and Bulbar Muscular Atrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBVS857X2202
Record Dates: First submitted 2013-12-29; First posted 2013-12-31 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Spinal and Bulbar Muscular Atrophy
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- BVS857 Part A Open label (Cohort 1) (Experimental): Participants received single doses of 0.01 mg/kg BVS857 intravenously (i.v.) on day 1, 0.01 mg/kg BVS857 subcutaneously (s.c.) on day 15, 0.03 mg/kg BVS857 s.c. on day 29, 0.06 mg/kg BVS857 s.c. on day 43 and 0.10 mg/kg BVS857 s.c. on day 57.
  Interventions: Drug: BVS857
- BVS857 Part A double blind (Cohort 2) (Experimental): Participants received single doses of 0.03 mg/kg BVS857 i.v on day 1, 0.03 mg/kg BVS857 s.c. on day 15, 0.06 mg/kg BVS857 s.c. on day 29, 0.10 mg/kg BVS857 s.c. on day 43 and 0.10 mg/kg BVS857 s.c. on day 57. (BVS857 concentrations differed on days 43 and 57.)
  Interventions: Drug: BVS857
- Placebo Part A double blind (Cohort 2) (Placebo Comparator): Participants received single doses of matching placebo i.v. on day 1 and matching placebo s.c. on days 15, 29, 43 and 57.
  Interventions: Drug: Placebo
- BVS857 Part B open-label (Cohort 4) (Experimental): Participants received 0.1 mg/kg BVS857 i.v. weekly for 12 weeks.
  Interventions: Drug: BVS857
- BVS857 Part B double blind (Cohort 5) (Experimental): Participants received 0.06 mg/kg (maximum 6 mg) BVS857 i.v. weekly for 12 weeks.
  Interventions: Drug: BVS857
- Placebo Part B double blind (Cohort 5) (Placebo Comparator): Participants received matching placebo i.v. to BVS857 weekly for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BVS857 — BVS857 lyophilisate in vial; the lyophilisate was reconstituted with sterile water for injection, diluted as appropriate, and administered either i.v. or s.c..
  Arms: BVS857 Part A Open label (Cohort 1); BVS857 Part A double blind (Cohort 2); BVS857 Part B double blind (Cohort 5); BVS857 Part B open-label (Cohort 4)
Drug: Placebo — Placebo lyophilisate in vial; the lyophilisate was reconstituted with sterile water for injection, diluted as appropriate, and administered either i.v. or s.c..
  Arms: Placebo Part A double blind (Cohort 2); Placebo Part B double blind (Cohort 5)

SUMMARY:
The purpose of this study was to determine if BVS857 is safe, tolerable and increases thigh muscle thickness in patients with spinal bulbar and muscular atrophy (SBMA).

ELIGIBILITY:
Key Inclusion Criteria:

* Genetic diagnosis of SBMA with symptomatic muscle weakness
* Able to complete 2 minute timed walk
* Serum IGF-1 level less than or equal to 170 ng/mL

Key Exclusion Criteria:

* Medically treated diabetes mellitus or known history of hypoglycemia
* History of Bell's palsy
* Treatment with systemic steroids > 10 mg/day (or equivalent dose); androgens or androgen reducing agents; systemic beta agonists; or other muscle anabolic drugs within the previous 3 months
* History of cancer, other than non-melanomatous skin cancer
* Retinopathy
* Papilledema Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2016-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (3):
  - Novartis Investigative Site, Orange, California
  - National Institutes of Health, Bethesda, Maryland
  - Novartis Investigative Site, Columbus, Ohio
- Novartis Investigative Site, Copenhagen, Denmark
- Novartis Investigative Site, Ulm, Germany
- Novartis Investigative Site, Padua, PD, Italy

REFERENCES:
- [Derived] Grunseich C, Miller R, Swan T, Glass DJ, El Mouelhi M, Fornaro M, Petricoul O, Vostiar I, Roubenoff R, Meriggioli MN, Kokkinis A, Guber RD, Budron MS, Vissing J, Soraru G, Mozaffar T, Ludolph A, Kissel JT, Fischbeck KH; BVS857 study group. Safety, tolerability, and preliminary efficacy of an IGF-1 mimetic in patients with spinal and bulbar muscular atrophy: a randomised, placebo-controlled trial. Lancet Neurol. 2018 Dec;17(12):1043-1052. doi: 10.1016/S1474-4422(18)30320-X. Epub 2018 Oct 15. PMID 30337273
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 2 parts, Part A and Part B. In Part A, Cohort 1 participants received open-label BVS857. Cohort 2 participants were randomized to double-blind BVS857 or double-blind placebo in a 2:1 ratio.
Pre-assignment Details: In Part B, Cohort 3 was not enrolled. Cohort 4 participants received open-label BVS857. Cohort 5 participants were randomized to double-blind BVS857 or double-blind placebo in a ratio of 18:10.
Groups:
- BVS857 Part A Double Blind (Cohort 2): Participants received single doses of 0.03 mg/kg BVS857 i.v. on day 1, 0.03 mg/kg BVS857 s.c. on day 15, 0.06 mg/kg BVS857 s.c. on day 29, 0.10 mg/kg BVS857 s.c. on day 43 and 0.10 mg/kg BVS857 s.c. on day 57. (BVS857 concentrations differed on days 43 and 57.)
Period: Overall Study
Arm/Group | BVS857 Part A Open Label (Cohort 1) | BVS857 Part A Double Blind (Cohort 2) | Placebo Part A Double Blind (Cohort 2) | BVS857 Part B Open-label (Cohort 4) | BVS857 Part B Double Blind (Cohort 5) | Placebo Part B Double Blind (Cohort 5)
Started | 2 | 4 | 2 | 2 | 18 | 9
Safety Analysis Set | 2 | 4 | 2 | 2 | 18 | 9
Pharmacokinetic (PK) Analysis Set | 2 | 4 | 0 | 2 | 18 | 0
Pharmacodynamic (PD) Analysis Set | 2 | 4 | 2 | 2 | 18 | 9
Completed | 0 | 1 | 2 | 0 | 16 | 9
Not Completed | 2 | 3 | 0 | 2 | 2 | 0
Not completed — Adverse Event | 2 | 3 | 0 | 0 | 2 | 0
Not completed — Abnormal laboratory value | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BVS857 Part A Open Label (Cohort 1) | BVS857 Part A Double Blind (Cohort 2) | Placebo Part A Double Blind (Cohort 2) | BVS857 Part B Open-label (Cohort 4) | BVS857 Part B Double Blind (Cohort 5) | Placebo Part B Double Blind (Cohort 5) | Total
Number analyzed (Participants) | 2 | 4 | 2 | 2 | 18 | 9 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.0 (5.66) | 56.0 (12.33) | 59.5 (7.78) | 41.5 (4.95) | 57.0 (55.5) | 54.0 (5.94) | 56.0 (10.33)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 2 | 4 | 2 | 2 | 18 | 9 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs), Serious Adverse Events (SAEs) and Deaths as a Measure of Safety and Tolerability
Description: Safety was monitored throughout the study.
Time Frame: After 78 days in Part A and after 85 days in Part B.
Population: The safety analysis set, which included participants who received any study drug, was analyzed.
Measure: Number; unit: Participants
Arm/Group | BVS857 Part A Open Label (Cohort 1) | BVS857 Part A Double Blind (Cohort 2) | Placebo Part A Double Blind (Cohort 2) | BVS857 Part B Open-label (Cohort 4) | BVS857 Part B Double Blind (Cohort 5) | Placebo Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 2 | 4 | 2 | 2 | 18 | 9
Participants
  Non-serious AEs | 2 | 4 | 2 | 1 | 17 | 8
  SAEs | 0 | 0 | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Mild, Moderate and Severe Adverse Events as a Measure of Safety and Tolerability
Description: Safety was monitored throughout the study.
Time Frame: After 78 days in Part A and after 85 days in Part B.
Population: The safety analysis set, which included participants who received any study drug, was analyzed.
Measure: Number; unit: Participants
Arm/Group | BVS857 Part A Open Label (Cohort 1) | BVS857 Part A Double Blind (Cohort 2) | Placebo Part A Double Blind (Cohort 2) | BVS857 Part B Open-label (Cohort 4) | BVS857 Part B Double Blind (Cohort 5) | Placebo Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 2 | 4 | 2 | 2 | 18 | 9
Participants
  Mild | 1 | 2 | 2 | 0 | 5 | 4
  Moderate | 1 | 2 | 0 | 0 | 11 | 3
  Severe | 0 | 0 | 0 | 0 | 1 | 1

3. Primary Outcome: Mean Percent Change From Baseline in Thigh Muscle Volume in Part B, Cohort 5
Description: Thigh muscle volume was assessed by magnetic resonance imaging (MRI). Change from baseline was calculated from the ratio of the post-baseline mean value to the baseline mean value: [(Day 85/baseline) - 1)] x 100. A positive change from baseline indicates improvement.
Time Frame: Baseline, Day 85
Population: The PD analysis set was considered for the analysis. However, only participants who had evaluable data at both baseline and day 85, were included in the analysis. The PD set included participants with evaluable PD data who received any study drug and had no protocol deviations with relevant impact on PD data.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | BVS857 Part B Double Blind (Cohort 5) | Placebo Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 15 | 9
Percent change | 0.0 (2.42) | -3.4 (4.79)
Statistical Analysis 1: Comparison: BVS857 Part B Double Blind (Cohort 5) vs Placebo Part B Double Blind (Cohort 5); Test type: Superiority or Other; p = 0.0164, ANCOVA; Geo-mean ratio = 1.037, 90% CI 2-sided [1.009 to 1.065]

4. Secondary Outcome: Mean Change From Baseline in Score on the Adult Myopathy Assessment Tool (AMAT) in Part B, Cohort 5
Description: The AMAT rated physical function and muscle endurance, with higher scores indicating better performance. The tool includes 7 timed functional tasks rated on a scale from 0 - 21 and 6 endurance tasks rated on a scale from 0 - 24. The range for the total score was from 0 (worst) to 45 (best). A positive change from baseline indicates improvement.
Time Frame: Baseline, Day 85
Population: The PD set included, which included participants with evaluable PD data who received any study drug and had no protocol deviations with relevant impact on PD data, was analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BVS857 Part B Double Blind (Cohort 5) | Placebo Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 18 | 9
score on a scale | 1.0 (4.20) | 2.3 (1.87)

5. Secondary Outcome: Mean Change From Baseline in Total Lean Body Mass (LBM) in Part B, Cohort 5
Description: LBM was assessed by dual-energy X-ray (DXA) absorptiometry. A positive change from baseline indicate improvement.
Time Frame: Baseline, Day 85
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | BVS857 Part B Double Blind (Cohort 5) | Placebo Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 17 | 8
kilograms | 0.77 (1.556) | 0.16 (1.199)

6. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: Observed Maximum Concentration Following Drug Administration (Cmax) in Part A, Cohort 1
Description: Serum samples were obtained for PK assessment.
Time Frame: Days 1, 15, 29, 43: pre-dose, 1, 4, 12, 24, 48, 168 hours post-dose
Population: For each time point, only participants from the PK set with valid measurements at that time point were analyzed. The PK analysis set included participants with at least one available valid PK concentration measurement who received any study drug and experienced no protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BVS857 Part A Open Label (Cohort 1)
Number analyzed (Participants) | 2
ng/mL
  Day 1, 0.01 mg/kg BVS857 i.v. | 184 (6.36)
  Day 15, 0.01 mg/kg BVS857 s.c. | 34.6 (48.9)
  Day 29, 0.03 mg/kg BVS857 s.c | 83.1 (20.3)
  Day 43, 0.06 mg/kg BVS857 s.c. | 74.2 (16.1)

7. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: Observed Maximum Concentration Following Drug Administration (Cmax) in Part A, Cohort 2
Description: Serum samples were obtained for PK assessment.
Time Frame: Days 1, 15, 29, 43: pre-dose, 1, 4, 12, 24, 48, 168 hours post-dose. Day 57: pre-dose, 1, 4, 12, 24, 48, 168, 504 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BVS857 Part A Double Blind (Cohort 2)
Number analyzed (Participants) | 4
ng/mL
  Day 1, 0.03 mg/kg BVS857 i.v. (n=4) | 393 (30.1)
  Day 15, 0.03 mg/kg BVS857 s.c. (n=3) | 77.3 (46.5)
  Day 29, 0.06 mg/kg BVS857 s.c. (n=2) | 113 (2.12)
  Day 43, 0.10 mg/kg BVS857 s.c. (n=3) | 191 (19.2)
  Day 57, 0.10 mg/kg BVS857 s.c. (n=1) | 232 (NA) — Standard deviation does not apply when n = 1.

8. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: Time to Reach the Maximum Concentration After Drug Administration (Tmax) in Part A, Cohort 1
Description: Serum samples were obtained for PK assessment.
Time Frame: Days 1, 15, 29, 43: pre-dose, 1, 4, 12, 24, 48, 168 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BVS857 Part A Open Label (Cohort 1)
Number analyzed (Participants) | 2
hours
  Day 1, 0.01 mg/kg BVS857 i.v. (n=2) | 4.04 (0.0566)
  Day 15, 0.01 mg/kg BVS857 s.c. (n=1) | 12.1 (NA) — Standard deviation does not apply when n = 1.
  Day 29, 0.03 mg/kg BVS857 s.c.(n=2) | 18.1 (8.41)
  Day 43, 0.06 mg/kg BVS857 s.c. (n=2) | 36.0 (16.8)

9. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: Time to Reach the Maximum Concentration After Drug Administration (Tmax) in Part A, Cohort 2
Description: Serum samples were obtained for PK assessment.
Time Frame: Day 1, 15, 29, 43: pre-dose, 1, 4, 12, 24, 48, 168 hours post-dose. Day 57: pre-dose, 1, 4, 12, 24, 48, 168, 504 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BVS857 Part A Double Blind (Cohort 2)
Number analyzed (Participants) | 4
hours
  Day 1, 0.03 mg/kg BVS857 i.v. (n=4) | 2.53 (1.70)
  Day 15, 0.03 mg/kg BVS857 s.c.(n=3) | 24.1 (0.100)
  Day 29, 0.06 mg/kg BVS857 s.c. (n=2) | 24.0 (0)
  Day 43, 0.10 mg/kg BVS857 s.c. (n=3) | 24.0 (0.200)
  Day 57, 0.10 mg/kg BVS857 s.c. (n=1) | 48.0 (NA) — Standard deviation does not apply when n = 1.

10. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: The Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) in Part A, Cohort 1
Description: Serum samples were obtained for PK assessment.
Time Frame: Days 1, 15, 29, 43: pre-dose, 1, 4, 12, 24, 48, 168 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | BVS857 Part A Open Label (Cohort 1)
Number analyzed (Participants) | 2
h*ng/mL
  Day 1, 0.01 mg/kg BVS857 i.v.(n=2) | 4630 (1200)
  Day 15, 0.01 mg/kg BVS857 s.c. (n=2) | 1060 (1500)
  Day 29, 0.03 mg/kg BVS857 s.c.(n=2) | 2720 (870)
  Day 43, 0.06 mg/kg BVS857 s.c.(n=2) | 5310 (4720)

11. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: The Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) in Part A, Cohort 2
Description: Serum samples were obtained for PK assessment.
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: H*ng/mL
Arm/Group | BVS857 Part A Double Blind (Cohort 2)
Number analyzed (Participants) | 4
H*ng/mL
  Day 1, 0.03 mg/kg BVS857 i.v.(n=4) | 9850 (4480)
  Day 15, 0.03 mg/kg BVS857 s.c. (n=3) | 6480 (5850)
  Day 29, 0.06 mg/kg BVS857 s.c. (n=2) | 7340 (5610)
  Day 43, 0.10 mg/kg BVS857 s.c. (n=3) | 14400 (3320)
  Day 57, 0.10 mg/kg BVS857 s.c. (n=1) | 28400 (NA) — Standard deviation does not apply when n = 1.

12. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: The Area Under the Plasma Concentration-time Curve From Zero to 48 Hours (AUC0_48h) in Part A, Cohort 1
Description: Serum samples were obtained for PK assessment.
Time Frame: Days 1, 15, 29, 43: pre-dose, 1, 4, 12, 24, 48, 168 hours post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | BVS857 Part A Open Label (Cohort 1)
Number analyzed (Participants) | 2
h*ng/mL
  Day 1, 0.01 mg/kg BVS857 i.v.(n=2) | 4620 (1200)
  Day 15, 0.01 mg/kg BVS857 s.c. (n=1) | 2120 (NA) — Standard deviation does not apply when n = 1.
  Day 29, 0.03 mg/kg BVS857 s.c. (n=2) | 2720 (870)
  Day 43, 0.06 mg/kg BVS857 s.c. (n=2) | 2210 (339)

13. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: The Area Under the Plasma Concentration-time Curve From Zero to 48 Hours (AUC0_48h) in Part A, Cohort 2
Description: Serum samples were obtained for PK assessment.
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | BVS857 Part A Double Blind (Cohort 2)
Number analyzed (Participants) | 4
h*ng/mL
  Day 1, 0.03 mg/kg BVS857 i.v. (n=4) | 7980 (1710)
  Day 15, 0.03 mg/kg BVS857 s.c. (n=3) | 2640 (1500)
  Day 29, 0.06 mg/kg BVS857 s.c. (n=2) | 3880 (735)
  Day 43, 0.10 mg/kg BVS857 s.c. (n=3) | 6390 (925)
  Day 57, 0.10 mg/kg BVS857 s.c. (n=1) | 7360 (NA) — Standard deviation does not apply when n = 1.

14. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: Observed Maximum Concentration Following Drug Administration (Cmax) in Part B, Cohort 4
Description: Serum samples were obtained for PK assessment.
Time Frame: Days 1: pre-dose, 1, 4, 24, 48 hours post-dose
Population: The PK analysis set, which included participants with at least one available valid PK concentration measurement who received any study drug and experienced no protocol deviations with relevant impact on PK data, was analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BVS857 Part B Open-label (Cohort 4)
Number analyzed (Participants) | 2
ng/mL | 2490 (799)

15. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: Observed Maximum Concentration Following Drug Administration (Cmax) in Part B, Cohort 5
Description: Serum samples were obtained for PK assessment.
Time Frame: Days 1 and 36: pre-dose, 1, 4, 24, 48 hours post-dose. Day 78: pre-dose, 1, 4, 24, 48, 168 hours post-dose.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BVS857 Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 18
ng/mL
  Day 1, 0.06 mg/kg BVS857 i.v. (n=18) | 854 (669)
  Day 36, 0.06 mg/kg BVS857 i.v. (n=16) | 790 (184)
  Day 78, 0.06 mg/kg BVS857 i.v. (n=16) | 712 (218)

16. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: Time to Reach the Maximum Concentration After Drug Administration (Tmax) in Part B, Cohort 4
Description: Serum samples were obtained for PK assessment.
Time Frame: Days 1: pre-dose, 1, 4, 24, 48 hours post-dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BVS857 Part B Open-label (Cohort 4)
Number analyzed (Participants) | 2
hours | 1.08 (0.0707)

17. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: Time to Reach the Maximum Concentration After Drug Administration (Tmax) in Part B, Cohort 5
Description: Serum samples were obtained for PK assessment.
Time Frame: Days 1 and 36: pre-dose, 1, 4, 24, 48 hours post-dose. Day 78: pre-dose, 1, 4, 24, 48, 168 hours post-dose.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BVS857 Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 18
hours
  Day 1, 0.06 mg/kg BVS857 i.v. (n=18) | 2.39 (1.54)
  Day 36, 0.06 mg/kg BVS857 i.v. (n=16) | 1.73 (1.20)
  Day 78, 0.06 mg/kg BVS857 i.v. (n=16) | 1.49 (1.04)

18. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: The Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) in Part B, Cohort 5
Description: Serum samples were obtained for PK assessment.
Time Frame: Day 36: pre-dose, 1, 4, 24, 48 hours post-dose. Day 78: pre-dose, 1, 4, 24, 48, 168 hours post-dose.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | BVS857 Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 18
h*ng/mL
  Day 36, 0.06 mg/kg BVS857 i.v. (n=1) | 13100 (NA) — Standard deviation does not apply when n = 1.
  Day 78, 0.06 mg/kg BVS857 i.v. (n=15) | 28000 (13500)

19. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857:The Area Under the Plasma Concentration-time Curve From Zero to 48 Hours (AUC0_48h) in Part B, Cohort 4
Description: Serum samples were obtained for the PK assessment.
Time Frame: Days 1: pre-dose, 1, 4, 24, 48 hours post-dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: H*ng/mL
Arm/Group | BVS857 Part B Open-label (Cohort 4)
Number analyzed (Participants) | 2
H*ng/mL | 40600 (1270)

20. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857:The Area Under the Plasma Concentration-time Curve From Zero to 48 Hours (AUC0_48h) in Part B, Cohort 5
Time Frame: Days 1 and 36: pre-dose, 1, 4, 24, 48 hours post-dose. Day 78: pre-dose, 1, 4, 24, 48, 168 hours post-dose.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | BVS857 Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 18
h*ng/mL
  Day 1, 0.06 mg/kg BVS857 i.v. (n=18) | 19400 (4160)
  Day 36, 0.06 mg/kg BVS857 i.v.(n=16) | 19600 (5240)
  Day 78, 0.06 mg/kg BVS857 i.v. (n=16) | 18100 (5850)

21. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: The Area Under the Serum Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau)
Description: Serum samples were obtained for PK assessment.
Time Frame: Part A: days 1, 15, 29, 43: pre-dose, 1, 4, 12, 24, 48, 168 hours post-dose. Day 57: pre-dose, 1, 4, 12, 24, 48, 168, 504 hours post-dose. Part B: days 1 and 36: pre-dose, 1, 4, 24, 48 hours post-dose. Day 78: pre-dose, 1, 4, 24, 48, 168 hours post-dose.
Population: This PK parameter was not analyzed in either Part A or Part B because there were insufficient data points after Cmax. Therefore, this parameter could not be calculated.
Arm/Group | BVS857 Part A Open Label (Cohort 1) | BVS857 Part A Double Blind (Cohort 2) | BVS857 Part B Open-label (Cohort 4) | BVS857 Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: The Terminal Elimination Half-life (T1/2)
Description: Serum samples were obtained for PK assessment.
Time Frame: as for outcome 21
Population: as for outcome 21
Arm/Group | BVS857 Part A Open Label (Cohort 1) | BVS857 Part A Double Blind (Cohort 2) | BVS857 Part B Open-label (Cohort 4) | BVS857 Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 0 | 0 | 0 | 0

23. Secondary Outcome: Plasma Pharmacokinetics (PK) of BVS857: The Area Under the Serum Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: Serum samples were obtained for PK assessment.
Time Frame: as for outcome 21
Population: as for outcome 21
Arm/Group | BVS857 Part A Open Label (Cohort 1) | BVS857 Part A Double Blind (Cohort 2) | BVS857 Part B Open-label (Cohort 4) | BVS857 Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 0 | 0 | 0 | 0

24. Secondary Outcome: Compare Dose Normalized Log-transformed AUCinf Following IV and SC Administrations
Description: Serum samples were obtained for PK assessment.
Time Frame: In Part A: days 1 and 15, pre-dose, 1, 4, 12, 24, 48, 168 hours post-dose.
Population: as for outcome 21
Arm/Group | BVS857 Part A Open Label (Cohort 1) | BVS857 Part A Double Blind (Cohort 2) | BVS857 Part B Open-label (Cohort 4) | BVS857 Part B Double Blind (Cohort 5)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | BVS857 Part A Open Label (Cohort 1) | Placebo Part A Double Blind (Cohort 2) | BVS857 Part A Double Blind (Cohort 2) | BVS857 Part B Open-label (Cohort 4) | BVS857 Part B Double Blind (Cohort 5) | Placebo Part B Double Blind (Cohort 5)
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/4 | 0/2 | 0/18 | 0/9
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 4/4 | 1/2 | 17/18 | 8/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BVS857 Part A Open Label (Cohort 1) (N=2) | Placebo Part A Double Blind (Cohort 2) (N=2) | BVS857 Part A Double Blind (Cohort 2) (N=4) | BVS857 Part B Open-label (Cohort 4) (N=2) | BVS857 Part B Double Blind (Cohort 5) (N=18) | Placebo Part B Double Blind (Cohort 5) (N=9)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eyelid haematoma (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Scleral hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Administration site hypersensitivity (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Catheter site extravasation (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infusion site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Infusion site pruritus (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 2 | 0 | 3 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Therapeutic response unexpected (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1 | 0 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Neutralising antibodies positive (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
Exostosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.